CLINICAL TRIAL: NCT02009683
Title: Multimodality Prediction of Success of Atrial Fibrillation Rhythm Control Strategy
Acronym: MULTI-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 13-2-033.3
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood biomarkers and SNPs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study the investigators aim to build a model to predict the maintenance of sinus rhythm (SR) after successful direct current cardioversion (DCC) incorporating standard predictors such as echocardiographic parameters, clinical parameter and 12-lead ECG parameters and new parameters, including 17-lead ECG, Oesophageal-ECG and single nucleotide polymorphisms (SNPs). Using this novel integrated prediction model will help in the identification of patients who will maintain SR after cardioversion. Another innovative aspect of our study is the use of daily rhythm monitoring using a versatile device (MyDiagnostick®). The clinical impact this study will have is that it helps the cardiologist to make a patient tailored strategy in the treatment of AF as advocated by the guidelines and to prevent exposing patients not likely to maintain SR to the potentially harmful side-effect of a rhythm-control strategy.

Primary objectives To show that a model incorporating the novel predictors 17-lead ECG, Oesophageal-ECG and SNPs is superior to existing models in predicting maintenance of sinus rhythm after successful DCC in patients with persistent AF.

Secondary objectives To assess the predictive value of new predictors (the Oesophageal-ECG, 17-lead ECG and SNPs) for maintenance of SR after successful DCC separately.

To assess the predictive value of new predictors (the Oesophageal-ECG, 17-lead ECG and SNPs) for time to recurrence of AF.

To assess the predictive value of predictors with respect to complete failure of cardioversion.

To assess the predictive value of predictors with respect to cardiovascular morbidity.

Hypothesis The investigators hypothesise that a model incorporating the novel predictors the 17-leads ECG, Oesophageal-ECG and SNPs performs significantly better than existing models using only clinical, echocardiographic and ECG parameters on a standard 12-lead ECG in predicting maintenance of SR after successful DCC. In addition the investigators hypothesise that Oesophageal-ECG is the best single predictor for maintenance of SR after successful DCC.

ELIGIBILITY:
Inclusion Criteria:

* Haemodynamic stable patients with persistent AF scheduled for DCC.
* Written informed consent.
* Patients > 18 years old.

Exclusion Criteria:

* Atrial flutter at time of DCC.
* Patients with known oesophageal disease.
* Patients with previous operations on throat or oesophagus.
* Postoperative atrial fibrillation.
* Patients with previous ablation for AF.
* Previous inclusion in this study.
* Patients on anti-arrhythmic drugs (AAD).
* Patients with pacemakers unable to detect AF and with a regular paced rhythm during AF.
* Planned ablation for AF.
* Myocardial infarction within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent atrial fibrillation scheduled for direct current cardioversion.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Maintenance of sinus rhythm after successful direct current cardioversion | 6 months

SECONDARY OUTCOMES:
Failure of direct current cardioversion | 1 day
Cardiovascular mortality | 6 months
Hospitalisation for cardiovascular events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: H Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands